CLINICAL TRIAL: NCT03229161
Title: Interval Walking Intervention for Pregnant Women Diagnosed With Gestational Diabetes Mellitus - a Pilot Study
Brief Title: Interval Walking Intervention for Pregnant Women Diagnosed With Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Danish Center for Strategic Research on Type 2 Diabetes (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Kathrine Kjaer, Principal investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CT20160156; S-20160156 (Other: The Regional Committees on Health Research Ethics for Southern Denmark); 16/40511 (Other: The Danish Data Protection Agency)
Record Dates: First submitted 2017-06-28; First posted 2017-07-25 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Intervention Model Description: This open-label randomized controlled trial aims to enroll 20 patients randomized (1:1) to a control- (Con) or IWT-group. Patients in both the IWT- and Con-group follows the standardized GDM care program for GDM patients at OUH through the 6-week intervention period, which consists of instruction of self-monitoring of BG levels, dietary guidance, and in some cases, insulin treatment. Additionally, the program also consists of close obstetric control visits and exercise guidance. All patients are instructed not to start any new type of PA after inclusion and continue their lives without any changes.
  Patients randomized to the IWT-group goes through a 6-week non-supervised IWT-program, where they are prescribed to conduct 3 IWT sessions per week of 40-50 minutes each.
  Before and after the 6-week intervention, maternal blood glucose (BG) levels is measured by continuous glucose monitoring, PA level measured using accelerometers and physical fitness measured using two walking tests.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IWT-group (Experimental): The IWT-group follows the standardized GDM care program for GDM patients at OUH and is prescribed to a 6-week non-supervised IWT-program consisting of 3 IWT sessions per week of 40-50 minutes each.
  Interventions: Behavioral: IWT-group
- Con-group (No Intervention): The con-group follows the standardized GDM care program for GDM patients at OUH

INTERVENTIONS:
Behavioral: IWT-group
  Arms: IWT-group

SUMMARY:
It is well-known that regular physical activity (PA) can improve glycemic control and physical fitness in type 2 diabetes patients. However, studies examining the effects of PA in patients with gestational diabetes mellitus (GDM) are limited. Interval walking training (IWT) is a careful type of PA consisting of repeatedly cycles of 3 min. fast and slow walking. The investigators aimed to examine, if IWT is feasible as PA intervention for GDM patients, and to examine the effects of IWT on glycemic control, PA levels and physical fitness.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM), defined as glucose intolerance and thus hyperglycemia with onset or first recognition during pregnancy, is steadily increasing in prevalence. In Denmark, the prevalence of GDM is around 2-3% of all pregnancies. GDM is associated with several adverse perinatal and maternal outcomes why early recognition and diagnosis is important. Early diagnosis and relevant treatment can prevent adverse outcomes of the baby and mother, such as macrosomia, shoulder dystocia, preeclampsia and hypoglycemia.

The glucose levels will often normalize shortly after birth; however, up to 50% of all women in Denmark diagnosed with GDM develop T2D during the first 10 years after the pregnancy, have a threefold risk of developing metabolic syndrome2 10, while the recurrence risk of developing GDM in subsequent pregnancies varies between 30-84%. Furthermore, long term increased risks for children born with macrosomia or by a mother with GDM include cardiovascular disease, obesity and T2D.

Glycemic control is a key factor in combatting the severe effects related to poorly controlled GDM. Management of GDM in Denmark consists of regular BG self-monitoring, dietary modifications, and in some cases insulin treatment. Additionally, obstetric control visits and PA advices are also a part of the standard GDM care program.

Compared to non-pregnant women, pregnant women must be more careful in relation to especially the type of PA, why supervised exercise is often recommended in order to ensure safe and correct guidance. This is a heavy economic burden, why a structured, non-supervised type of PA with low a risk of injury, possibly high compliance and continuous monitoring would be preferable. Interval walking training (IWT) is a lenient type of structured, non-supervised PA. This type of PA is associated with an improved glucose regulation in patients with T2D after 4 months of IWT 5 times weekly (60 min./session) (Karstoft et al., 2013). Due to similar metabolic dysregulations in patients with T2D and GDM, the investigators are apt to believe that IWT, if feasible, can improve glycemic control in GDM patients. Furthermore, it is obvious to believe that IWT can be implemented as regular PA in GDM patients, as one study has shown that pregnant women mostly prefer walking as a type of PA during pregnancy.

This open-label randomized controlled trial aims to enroll 20 patients randomized (1:1) to a control- (Con) or IWT-group. Both groups will follow the standard GDM care program at Odense University Hospital. Additionally, the IWT-group is prescribed three weekly IWT sessions of 40-50 minutes each for 6 weeks. Each IWT session is guided and controlled by the smartphone application 'InterWalk', which individualize the training intensity to current fitness level of the patient through an on-board fitness test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with GDM by a 2 hour oral glucose tolerance test with a BG level of >9.00mmol/l at 2 hours
* Danish speaking
* >18 years of age
* Live <20 kilometers from Odense city center

Exclusion Criteria:

* Pelvic pains
* Untreated depression
* Walking disabilities
* Pregnancy-related complications
* >32 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As only women can be diagnosed with gestational diabetes mellitus, only women are eligible in participating in the study.
Enrollment: 3 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Compliance to the prescribed IWT-intervention | After the 6-week intervention period
  Compliance defined as adherence to the prescribed IWT-intervention
Compliance to the prescribed IWT-intervention | After the 6-week intervention period
  Compliance defined as the quality of the the IWT sessions

SECONDARY OUTCOMES:
Glycemic control | Before and after the 6-week intervention period
  Blood glucose variations measured by 48-hour continuous glucose monitoring
Physical activity level | 7 days before and after the 6-week intervention period, and the first and last 5 days during the 6-week intervention period
  Physical activity level measured by accelerometers
Physical fitness | Before and after the 6-week intervention period
  Physical fitness measured by the on-board fitness test in the InterWalk application and a 6-minute walking test

OTHER OUTCOMES:
Blood pressure | Before and after the 6-week intervention period
  30 minutes systolic and diastolic Blood Pressure (BP) together with pulse wave velocity (PWV) was measured by using the Mobil-O Graph® PWA device. BP and PWV was measured every 3 minutes for 30 minutes in a sitting position with the assessor only being in the room during the first measurement to ensure adequate quality.
Physical and mental health | Before and after the 6-week intervention period
  Perceived physical and mental health was measured using the SF-12 questionnaire.
BMI | Before and after the 6-week intervention period
  Body height and body weight were objectively measured. Height was measured in an upright standing position without shoes by using a stadiometer. Weight was also measured in a standing position without shoes by using a digital scale. Height and weight was measured to the nearest 0.5 centimeter and 0.1 kilo respectively. BMI was calculated based on measured height and weight

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Centre of strategic research of type 2 diabetes, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No